CLINICAL TRIAL: NCT07008287
Title: A Multicenter, Non-interventional, Observational Study of Taletrectinib for Advanced ROS1+ NSCLC With Brain Metastases
Brief Title: Real-world Study of Taletrectinib for Advanced ROS1+ NSCLC With Brain Metastases
Status: Recruiting | Type: Observational
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: IBI344-RWS-002
Record Dates: First submitted 2025-05-28; First posted 2025-06-06 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — taletrectinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cohort 1: ROS1 fusion positive NSCLC patients with brain metastases who received taletrecitnib
  Interventions: Drug: Taletrectinib

INTERVENTIONS:
Drug: Taletrectinib — Taletrectinib, 600mg, QD
  Other Names: AB-106; DS-6051b

SUMMARY:
This is a multicenter, non-interventional, observational real-world study to evaluate the efficacy and safety of Taletrectinib in ROS1-positive non-small cell lung cancer (NSCLC) with brain metastases. Patients deemed eligible for Taletrectinib by their physicians were enrolled after providing informed consent. Taletrectinib will be administered according to clinical practice and data on treatment patterns, clinical outcomes, and safety will be collected during routine evaluations.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following criteria to be eligible for enrollment into the study:

1. Age ≥ 18 years.
2. Histologically or cytologically metastatic NSCLC (UICC/AJCC TNM Staging System, 9th Edition, Stage Ⅳ).
3. At least one measurable target tumor lesion as accessed by RECIST v1.1 criteria.
4. Radiographically confirmed brain metastasis(es) , with stable CNS symptoms within 2 weeks prior to enrollment.
5. Documented ROS1 gene fusion identified by an approved molecular testing method (FISH, RT-PCR, or NGS).
6. Considered by the investigator to be candidates for Taletrectinib treatment ; OR Patients with ≤6 months of prior Taletrectinib exposure enrolled retrospectively. (Note: For retrospective patients deceased before enrollment, waiver of informed consent is required. Patients who initiated and discontinued treatment within 6 months prior to signing informed consent are eligible).
7. Signed Informed Consent.

Exclusion Criteria:

Patient presenting with any of the following criteria will not be included in the study：

1. Patients with driver gene mutations/alterations that have approved targeted therapies , including but not limited to EGFR, ALK, RET, etc.
2. Currently participating in other interventional clinical trials or having received investigational drug treatment within 4 weeks prior to enrollment .
3. Pregnancy or breastfeeding.
4. Patients with uncontrolled co-morbidities who are assessed by the investigator not to receive targeted therapy.
5. Other conditions that are assessed by the investigator to be unsuitable for enrollment in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ROS1-positive non-small cell lung cancer (NSCLC) with brain metastasis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
ORR | 6 months
  Objective response rate
iORR | 6 months
  Intracranial objective response rate

SECONDARY OUTCOMES:
PFS | 25 months
  Progression free survival
DoR | 25 months
  Duration of response
DCR | 6 months
  Disease control rate
OS | 51 months
  Overall survival
iPFS | 25 months
  Intracranial progress free survival
iDoR | 6 months
  Intracranial duration of response
iDCR | 6 months
  Intracranial disease control rate
Adverse events | 25 months
  Type, incidence, severity, timing, seriousness, and relatedness of adverse events and laboratory abnormalities, graded by the NCI CTCAE 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No